CLINICAL TRIAL: NCT03621020
Title: Clinical Performance Evaluation of T-TAS 01 PL Chip
Status: Completed | Type: Observational
Sponsor: Hikari Dx, Inc. (Other)
Collaborators: Fujimori Kogyo Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: TQPL-RD-121-1
Record Dates: First submitted 2018-08-05; First posted 2018-08-08 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Platelet Dysfunction; Von Willebrand Diseases; Healthy; Congenital Platelets Abnormality
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (5):
- Healthy controls: Subjects not taking medications with antiplatelet effects, without evidence of vWD or history of congenital platelet abnormalities, without history of significant bleeding.
  Interventions: Diagnostic Test: T-TAS 01 PL Chip; Diagnostic Test: PFA-100 Col/Epi and Col/ADP
- Aspirin monotherapy: Subjects taking 81+ mg daily aspirin and no additional medications with antiplatelet effects, without evidence of vWD or history of congenital platelet abnormalities, without history of significant bleeding.
  Interventions: Diagnostic Test: T-TAS 01 PL Chip; Diagnostic Test: PFA-100 Col/Epi and Col/ADP
- von Willebrand Disease: Subjects diagnosed with vWD (all types except Type 2N), not taking medications with antiplatelet effects, and history of clinically significant bleeding.
  Interventions: Diagnostic Test: T-TAS 01 PL Chip; Diagnostic Test: PFA-100 Col/Epi and Col/ADP
- Glanzmann's Thrombasthenia: Subjects diagnosed with Glanzmann's Thrombasthenia, not taking medications with antiplatelet effects, and history of clinically significant bleeding.
  Interventions: Diagnostic Test: T-TAS 01 PL Chip; Diagnostic Test: PFA-100 Col/Epi and Col/ADP
- Dual antiplatelet therapy (DAPT): Subjects taking 81 mg daily aspirin and either 75 mg daily clopidogrel, 10 mg daily prasugrel, or 180 mg daily ticagrelor
  Interventions: Diagnostic Test: T-TAS 01 PL Chip

INTERVENTIONS:
Diagnostic Test: T-TAS 01 PL Chip — Flow chamber microchip system specific for measuring primary hemostatic ability
Diagnostic Test: PFA-100 Col/Epi and Col/ADP — System for measuring platelet dysfunction
  Groups: Aspirin monotherapy; Glanzmann's Thrombasthenia; Healthy controls; von Willebrand Disease

SUMMARY:
This study will measure primary hemostatic ability using the T-TAS 01 System with PL chip, with a comparison to clinical truth.

DETAILED DESCRIPTION:
This study will measure primary hemostatic ability using the T-TAS 01 System with PL chip, with a comparison to clinical truth. The study will be conducted at 3 locations in the United States and will enroll approximately 335 subjects. The following subject populations will be enrolled into the study (expected enrollment numbers indicated in parentheses):

* Ostensibly healthy subjects without primary hemostasis abnormalities, e.g. a "healthy platelet" normal control population (N = 150)
* Subjects taking 81+ mg daily aspirin (N = 81)
* Subjects taking dual antiplatelet therapy (N = 51)
* Subjects with von Willebrand disease (vWD; N = 47)
* Subjects with Glanzmann's thrombasthenia (N = 5)

Subjects may be recruited either prospectively or based on their simultaneous participation in other studies involving blood collection, provided that the enrollment criteria. Blood samples will be collected after enrollment and subject participation will be complete after blood samples are collected and all necessary information is collected to complete the case report form (CRF). Blood sample testing with T-TAS 01 will occur locally at each investigational site. Blood sample testing for clinical truth assessment may be tested either locally or remotely, depending on the local availability of the various tests used for determining clinical truth.

ELIGIBILITY:
Normal Controls:

Inclusion Criteria

* Males and females age 21 years or older.
* Able and willing to provide written informed consent. Exclusion Criteria
* Abnormal results from assays used to establish clinical truth (retrospective exclusion).
* Hospitalization or doctor's visits within prior 30 days, except for routine checkup/physical examination.
* Use of antiplatelet therapy within the past 14 days, e.g. aspirin, clopidogrel, prasugrel, ticagrelor, cilostazol.
* Use of anticoagulant drugs within the past 14 days, e.g. heparin, bivalirudin, warfarin, rivaroxaban, and apixaban.
* Use of certain nonsteroidal anti-inflammatory drugs (NSAIDs) such as celecoxib, rofecoxib, etc. within the past 14 days.
* History of anemia.
* Known thrombocytopenia (platelet count < 100,000/μL).
* Significant renal dysfunction or dialysis.
* History of platelet disorders e.g. von Willebrand factor deficiency, Glanzmann's thrombasthenia or Bernard-Soulier syndrome.
* History of hemophilia or bleeding disorders.
* History of bleeding, with Bleeding Score ≥ 5 (Tosetto J Thromb Haemost 2006). See Appendix A. Scores will be assigned based on health history according to the following categories:

  * Epistaxis
  * Cutaneous bleeding
  * Bleeding from minor wounds
  * Bleeding from oral cavity
  * Gastrointestinal bleeding
  * Bleeding from tooth extraction
  * Surgical bleeding
  * Menorrhagia
  * Post-partum hemorrhage
  * Muscle hematoma
  * Hemarthrosis
  * Central nervous system bleeding
* Females who are in the last trimester of pregnancy, or are breastfeeding.
* Known active gastrointestinal disease including peptic ulcers, gastro-esophageal reflux disease (GERD), and hyperacidity.
* Currently participating in a study involving an investigational drug or compound known to affect coagulation or hemostasis.
* Subjects with significant past medical history as determined by the Investigator that would pose safety concerns or interfere with the study goals.

Antiplatelet Therapy Subjects:

Inclusion Criteria

* Males and females age 21 years or older.
* Continuous daily ingestion of one of the following antiplatelet therapy regimens:

  * 81 mg or higher aspirin
  * 81 mg or higher aspirin plus 75 mg daily clopidogrel
  * 81 mg or higher aspirin plus 10 mg daily prasugrel
  * 81 mg aspirin plus 180 mg daily ticagrelor
* Able and willing to provide written informed consent. Exclusion Criteria
* Use of antiplatelet therapy besides aspirin (e.g. clopidogrel, prasugrel, ticagrelor, cilostazol, abciximab, eptifibatide) within the past 14 days.
* Use of anticoagulant drugs within the past 14 days, e.g. heparin, bivalirudin, warfarin, rivaroxaban, and apixaban.
* Use of certain nonsteroidal anti-inflammatory drugs (NSAIDs) such as celecoxib, rofecoxib, etc. within the past 14 days.
* Significant renal dysfunction or dialysis.
* Known thrombocytopenia (platelet count < 100,000/μL).
* History of platelet disorders e.g. von Willebrand factor deficiency, Glanzmann thrombasthenia or Bernard-Soulier syndrome.
* History of hemophilia or bleeding disorders.
* Females who are in the last trimester of pregnancy, or are breastfeeding.
* Known active gastrointestinal disease including peptic ulcers, gastro-esophageal reflux disease (GERD), and hyperacidity.
* Currently participating in a study involving an investigational drug or compound known to affect coagulation or hemostasis.
* Subjects with significant past medical history as determined by the Investigator that would pose safety concerns or interfere with the study goals.

vWD Subjects: Inclusion Criteria

* Males and females age 21 years or older.
* Prior diagnosis of von Willebrand disease type 1, 2A, 2B, 2M, or 3
* History of bleeding, with Bleeding Score ≥ 5, which is 99% specific for vWD (Tosetto J Thromb Haemost 2006). See Appendix A. Scores will be assigned based on health history according to the following categories:

  * Epistaxis
  * Cutaneous bleeding
  * Bleeding from minor wounds
  * Bleeding from oral cavity
  * Gastrointestinal bleeding
  * Bleeding from tooth extraction
  * Surgical bleeding
  * Menorrhagia
  * Post-partum hemorrhage
  * Muscle hematoma
  * Hemarthrosis
  * Central nervous system bleeding
* Able and willing to provide written informed consent. Exclusion Criteria
* Prior diagnosis of von Willebrand disease type 2N
* Receiving desmopressin or vWF replacement therapy within the past 2 weeks.
* Use of antiplatelet therapy within the past 14 days.
* Use of anticoagulant drugs within the past 14 days, e.g. heparin, bivalirudin, warfarin, rivaroxaban, and apixaban.
* Use of certain nonsteroidal anti-inflammatory drugs (NSAIDs) such as celecoxib, rofecoxib, etc. within the past 14 days.
* Significant renal dysfunction or dialysis.
* Known thrombocytopenia (platelet count < 100,000/μL).
* Females who are in the last trimester of pregnancy, or are breastfeeding.
* Currently participating in a study involving an investigational drug or compound known to affect coagulation or hemostasis.
* Subjects with significant past medical history as determined by the Investigator that would pose safety concerns or interfere with the study goals.

Glanzmann's Thrombasthenia Subjects:

Inclusion Criteria

* Males and females age 21 years or older.
* Prior diagnosis of Glanzmann's thrombasthenia
* History of bleeding.
* Able and willing to provide written informed consent. Exclusion Criteria
* Use of antiplatelet therapy within the past 14 days.
* Use of anticoagulant drugs within the past 14 days, e.g. heparin, bivalirudin, warfarin, rivaroxaban, and apixaban.
* Use of certain nonsteroidal anti-inflammatory drugs (NSAIDs) such as celecoxib, rofecoxib, etc. within the past 14 days.
* Significant renal dysfunction or dialysis.
* Known thrombocytopenia (platelet count < 100,000/μL).
* Females who are in the last trimester of pregnancy, or are breastfeeding.
* Currently participating in a study involving an investigational drug or compound known to affect coagulation or hemostasis.
* Subjects with significant past medical history as determined by the Investigator that would pose safety concerns or interfere with the study goals.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ostensibly healthy subjects without primary hemostasis abnormalities, e.g. a "healthy platelet" normal control population Subjects taking 81+ mg daily aspirin Subjects taking dual antiplatelet therapy Subjects with von Willebrand disease (vWD) Subjects with Glanzmann's thrombasthenia
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity for detecting defects in primary hemostasis | Baseline
  Sensitivity and specificity of the T-TAS 01 PL chip assay against clinical truth

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Dahlen, Ph.D., Study Director — Hikari Dx, Inc.
Locations (6):
- United States (5):
  - San Francisco General Hospital, San Francisco, California
  - University of Iowa, Iowa City, Iowa
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Inova Cardiology Baltimore, Lutherville, Maryland
  - Inova Heart and Vascular Institute, Falls Church, Virginia
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, CA, France

IPD SHARING:
Plan to Share IPD: No